CLINICAL TRIAL: NCT05405790
Title: Antibiotic Prophylaxis for Thoracic EndoVascular Aortic Repair
Brief Title: Antibiotic Prophylaxis for TEVAR
Status: Terminated | Type: Observational
Why Stopped: Unable to enroll a sufficient number of patients
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hongkun Zhang, MD, Head of Vascular Surgery, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20220172A
Record Dates: First submitted 2022-05-30; First posted 2022-06-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Aortic Dissection; Aortic Diseases; Aortic Aneurysm, Thoracic; Coarctation of Aorta; Hematoma; Aorta
Keywords: Antibiotic prophylaxis; TEVAR; Fever; MAGIC classification
MeSH Terms: conditions — Aortic Dissection; Aortic Diseases; Aortic Aneurysm, Thoracic; Aortic Coarctation; Hematoma; Fever | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients receiving TEVAR
  Interventions: Procedure: thoracic endovascular aortic repair

INTERVENTIONS:
Procedure: thoracic endovascular aortic repair — In The TEVAR procedure, we implant a stent graft into the diseased area of the thoracic artery, providing a route for the blood to flow within the stent graft and excluding the diseased aorta.

SUMMARY:
The infection rate of thoracic endovascular aortic repair (TEVAR) is unknown due to a lack of epidemiological data. The rate currently available comes from researches conducted decades ago, when open surgery was the standard of care. Because of the potentially fatal consequences of a stent graft infection in the thoracic aorta, the investigators tend to prescribe antibiotic prophylaxis for at least three days. In this study, the investigators are going to collect data on patients receiving TEVAR in the past five years and provide the following information: a. the infection rate (MAGIC classification), b. the rate of fever, c. the results of the lab tests, such as the WBC count and C-reaction protein. d. risk factors associated with infection and fever.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with thoracic aortic diseases
2. Received TEVAR

Exclusion Criteria:

1. Suspected infectious aortic disease, such as a mycotic aneurysm.
2. TEVAR combined with open surgery
3. Antibiotics have been used more than 24 hours before the operation
4. Combined with immune deficiency disease or using hormone or immunosuppressant；
5. The treatment is for the complications of TEVAR, such as endoleak
6. Endovascular aortic repair for abdominal aortic disease
7. History of open aortic surgery or heart surgery.
8. Revascularization of visceral arteries during the TEVAR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with thoracic aortic dissection, thoracic aortic aneurysm, thoracic aortic intramural hematoma, or other thoracic aortic diseases and underwent TEVAR during hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Infection rate after TEVAR | during hospitalization (up to post-operation day 14)
  Infection rate via MAGIC classification
Infection rate at one month after TEVAR | One month after TEVAR
  Infection rate via MAGIC classification
Infection rate at six months after TEVAR | Six months after TEVAR
  Infection rate via MAGIC classification
Infection rate at one year after TEVAR | One year after TEVAR
  Infection rate via MAGIC classification

SECONDARY OUTCOMES:
Fever | one day, two days, three days, one month, six months, one year after TEVAR
  Defined as temperature ≥38.5℃
WBC count | one day, two days, three days after TEVAR
C-reaction protein | one day after TEVAR

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided